CLINICAL TRIAL: NCT03779945
Title: Application of Platelet-Rich-Plasma in Posterolateral Lumbar Fusion
Brief Title: Effect of Platelet-Rich-Plasma in Spine Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Micheal Bassem Elia, orthopedics resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRP in lumbar fusion
Record Dates: First submitted 2018-05-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Platelet-Rich Plasma
Keywords: PRP

STUDY DESIGN:
Intervention Model Description: single center, prospective randomized comparative trial
Who Masked: Outcomes Assessor
Masking Description: the person performing the statistical analysis shall be masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- posteriolateral lumbar fusion +bone graft+ PRP (Active Comparator): the addition of autologous platelet rich plasma to the bone graft
  Interventions: Biological: autologous platelet rich plasma
- posteriolateral lumbar fusion+bone graft only (Active Comparator): posteriolateral lumbar fusion with adding autologus bone graft alone posteriolateral lumbar fusion only
  Interventions: Procedure: posteriolateral lumbar fusion only

INTERVENTIONS:
Biological: autologous platelet rich plasma — adding autologous platelet rich plasma to the bone graft harvested from the patient
  Arms: posteriolateral lumbar fusion +bone graft+ PRP
Procedure: posteriolateral lumbar fusion only — performing posteriolateral lumbar fusion without using platelet rich plasma
  Arms: posteriolateral lumbar fusion+bone graft only

SUMMARY:
The objective of this study is to evaluate the fusion rate after the use of platelet rich plasma with autolgus bone graft and comparing it with bone graft alone

DETAILED DESCRIPTION:
The study will be submitted for approval by the Ethics Committee of Faculty of Medicine, Assiut University, and written informed consent will be obtained from all patients prior to enrollment. The study population will be selected from patients attending the Department of Orthopedics and Trauma surgery, Assiut University hospitals.

A total of 104 patients treated with single level degenerative or lytic lumbar Spondylolisthesis indicated for PLF will be included ,patients will be classified into 2 groups Group A:Of 52 patients PLF + autologus bone graft+ PRP Group B: Of 52 patients treated with PLF + autologus bone graft only without adding PRP

Methods of evaluation

* History taking.
* Full clinical and neurological examination
* Radiological evaluation by x-ray (antero posterior, lateral, and, CT scans provide excellent views of bony detail) and MRI if needed Method of randomization By shuffling cards method the candidate patient will choose one card from104 cards 52 of them containing fusion with PRP and the other 52 contaning Fusion without PRP

Platelet-rich plasma (PRP is obtained using a two-stage centrifugation process:

Whole blood sample will be drawn from the participant and be collected in a sterile tube containing anticoagulant (sodium citrate 3.8% or Ethylenediaminetetra acetic acid). The tube will be centrifuged at 160xg relative centrifugal force (about 1000 round per minute) for 10 min in a centrifugal apparatus. The first spin will separate platelet poor plasma at the top from red blood cells at the bottom and platelet rich plasma above (mixed with the white blood cells in the buffy coat). The Platelet poor plasma, Platelet rich plasma and a few red blood cells will be aspirated into a new tube, mixed and in the second spin, the tube will be centrifuged at 400xg relative centrifugal form (about 1500 round per minute) for another 10 minutes. The upper section will consist of Platelet poor plasma and the Platelet rich plasma will be collected at the bottom of the tube in the form of pellet. Then, Platelet poor plasma and Platelet rich plasma will be aspirated and mixed (discarding the upper portion). Prior to treatment calcium chloride 3% will be added to activate platelets specimen

ELIGIBILITY:
Inclusion Criteria:

degenerative or lytic Spondylolisthesis.

Degenerative disc disease requiring posterior lumbar fusion not responding to medical treatment for 1 year.

Age between 20 & 75 years.

Single level fusion

Exclusion Criteria:

Multiple levels patient Traumatic Spondylolisthesis Previous lumbar spine surgery. Other lumbar spine pathology severe osteoporosis Patients younger than 20 years old. Patients older than 75 years old. Immunocompromised patients (eg. Chronic renal failure)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-20 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-01-20 (Estimated)

PRIMARY OUTCOMES:
Lenke classiﬁcation of posterolateral fusion success | 6 month to1 year post-operative
  the degree of bridging bone across the fused vertebral bodies by using xray and CT scan

SECONDARY OUTCOMES:
modified Oswestry disability index , | 6 month to 1 year post-operative
  the functional outcome on the patient
visual analogue scale | 6 month to 1 year post-operative
  the amount of pain sensed by the patient pre and post-operative

CONTACTS AND LOCATIONS:
Overall Officials: El Moataz A Zohny El Sabrout, professor, Study Chair — Assiut University; Essam M Abdelmoneim Elmorshedy, Lecturer, Principal Investigator — Assiut University; . Belal O Mohamed Elnady, Lecturer, Principal Investigator — Assiut University

REFERENCES:
- [Background] Kubota G, Kamoda H, Orita S, Yamauchi K, Sakuma Y, Oikawa Y, Inage K, Sainoh T, Sato J, Ito M, Yamashita M, Nakamura J, Suzuki T, Takahashi K, Ohtori S. Platelet-rich plasma enhances bone union in posterolateral lumbar fusion: A prospective randomized controlled trial. Spine J. 2019 Feb;19(2):e34-e40. doi: 10.1016/j.spinee.2017.07.167. Epub 2017 Jul 20. PMID 28735763
- [Background] Shiga Y, Orita S, Kubota G, Kamoda H, Yamashita M, Matsuura Y, Yamauchi K, Eguchi Y, Suzuki M, Inage K, Sainoh T, Sato J, Fujimoto K, Abe K, Kanamoto H, Inoue M, Kinoshita H, Aoki Y, Toyone T, Furuya T, Koda M, Takahashi K, Ohtori S. Freeze-Dried Platelet-Rich Plasma Accelerates Bone Union with Adequate Rigidity in Posterolateral Lumbar Fusion Surgery Model in Rats. Sci Rep. 2016 Nov 11;6:36715. doi: 10.1038/srep36715. PMID 27833116
- [Background] Imagama S, Ando K, Kobayashi K, Ishikawa Y, Nakamura H, Hida T, Ito K, Tsushima M, Matsumoto A, Morozumi M, Tanaka S, Machino M, Ota K, Nakashima H, Takamatsu J, Matsushita T, Nishida Y, Ishiguro N, Matsuyama Y. Efficacy of Early Fusion With Local Bone Graft and Platelet-Rich Plasma in Lumbar Spinal Fusion Surgery Followed Over 10 Years. Global Spine J. 2017 Dec;7(8):749-755. doi: 10.1177/2192568217696690. Epub 2017 Apr 11. PMID 29238638
- [Background] Tarantino R, Donnarumma P, Mancarella C, Rullo M, Ferrazza G, Barrella G, Martini S, Delfini R. Posterolateral arthrodesis in lumbar spine surgery using autologous platelet-rich plasma and cancellous bone substitute: an osteoinductive and osteoconductive effect. Global Spine J. 2014 Aug;4(3):137-42. doi: 10.1055/s-0034-1376157. Epub 2014 May 3. PMID 25083353